CLINICAL TRIAL: NCT04604769
Title: Perceived Stress and Needs Among Medical Staff in ICU During COVID-19 Crisis
Brief Title: Perceived Stress Among ICU Medical Staff During COVID-19 Crisis
Acronym: ICUcovid
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Audrey Vanhaudenhuyse, PhD, Head of the Sensation and Perception Research Group, GIGA Consciouness, University of Liege
Other Study IDs: stressICUcovid
Record Dates: First submitted 2020-04-27; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Coronavirus; Nurse's Role; Professional Stress
Keywords: coronavirus; covid-19; pandemia; professional stress; burnout; nursing; intensive care units (ICU); infection; work organization
MeSH Terms: conditions — Coronavirus Infections; Occupational Stress; COVID-19; Burnout, Psychological; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Daily routine, control group: ICU medical staff were asked about their stress and causes of stress during their daily professional life.
- During Covid-19: ICU medical staff were asked about their stress and causes of stress in their daily professional life during COVID-19 crisis.

SUMMARY:
The objective of this study is to compare psychological distress and needs of nurses in ICU before and during coronavirus pandemic.

DETAILED DESCRIPTION:
Well-being of caregivers and stress management in intensive care units are essential keys to an adequate quality of care, especially during the anxious context of coronavirus pandemic. Taking care of numerous patients, the increasing work and mental charges, facing death, the need of material and changes in work organization are all elements that can influence stress among medical workers. Considering real causes of stress and what are the needs of the medical team is fundamental for developing concrete actions to ease the workloads. A few studies were conducted in China on psychological distress of medical staff during COVID-19. According to these few studies about psychological distress in ICU, investigators think that stress scores during COVID-19 could be increased among nurses during pandemic. The second hypothesis is that causes of stress would be not so different from normal care but could be amplified by the actual situation. One point to take into consideration is that most of the studies were conducted in China and medical policy and hospital organization are different in Belgium. The objective of the study is to compare psychological distress and needs of nurses in ICU before and during coronavirus pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years old
* working in ICU for at least November 2019
* working in ICU regularly since March 2020
* Medical and paramedical professionals
* Working in direct contact with COVID patients

Exclusion Criteria:

* Medical professionals from others departments
* Internship students
* External volunteers for COVID
* Non front-line nurses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurses and doctors working in intensive care units before and during the COVID pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
stress at work | change from baseline at one year
  Job Content Questionnaire (Karasek, 1979)
stress in a medical unit | change from baseline at one year
  Nursing Stress Questionnaire (Gray-Toft, 1981)

SECONDARY OUTCOMES:
hobby activities | change from baseline at one year
  We will ask if they are used to do activities like hypnosis, yoga, mediation, sport, etc. This factor could help us to know if these activities can help and if we have to promote them in the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie Nyssen, Principal Investigator — Université de Liège
Locations (1):
- University of Liège, Liège, Province De Liège, Belgium